CLINICAL TRIAL: NCT06079268
Title: Assessment of the Diagnostic Performance of Qualitative Ultrasound Assessment of Gastric Contents for the Detection of Gastric Fluid Volume ≥ 1.25 ml/kg in Children
Brief Title: Diagnostic Performance of Gastric Ultrasound in Children
Acronym: QUALIGASTR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 69HCL23_0690
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 0 ml/kg of water (Experimental): The child does not drink water, and then the gastric ultrasound is performed 3 minutes later blindly to the ingested volume.
  Interventions: Other: the initial gastric ultrasound; Other: the gastric ultrasound last 3 minutes
- 0.6 ml/kg of water (Experimental): The child drinks 0.6 ml/kg water, and then the gastric ultrasound is performed 3 minutes later blindly to the ingested volume.
  Interventions: Other: the initial gastric ultrasound; Other: the gastric ultrasound last 3 minutes
- 1 ml/kg of water (Experimental): The child drinks 1 ml/kg water, and then the gastric ultrasound is performed 3 minutes later blindly to the ingested volume.
  Interventions: Other: the initial gastric ultrasound; Other: the gastric ultrasound last 3 minutes
- 1.25 ml/kg of water (Experimental): The child drinks 1.25 ml/kg water, and then the gastric ultrasound is performed 3 minutes later blindly to the ingested volume
  Interventions: Other: the initial gastric ultrasound; Other: the gastric ultrasound last 3 minutes
- 1.5 ml/kg of water (Experimental): The child drinks 1.5 ml/kg water, and then the gastric ultrasound is performed 3 minutes later blindly to the ingested volume.
  Interventions: Other: the initial gastric ultrasound; Other: the gastric ultrasound last 3 minutes
- 2 ml/kg of water (Experimental): The child drinks 2 ml/kg water, and then the gastric ultrasound is performed 3 minutes later blindly to the ingested volume.
  Interventions: Other: the initial gastric ultrasound; Other: the gastric ultrasound last 3 minutes

INTERVENTIONS:
Other: the initial gastric ultrasound — Non-invasive gastric antrum ultrasound examinations will utilize a probe with a frequency of 2-5.5 MHz and a linear probe with a frequency of 10 MHz, enabling the evaluation of the gastric antrum's appearance
Other: the gastric ultrasound last 3 minutes — Non-invasive gastric antrum ultrasound examinations will utilize a probe with a frequency of 2-5.5 MHz and a linear probe with a frequency of 10 MHz, enabling the evaluation of the gastric antrum's appearance

SUMMARY:
Pulmonary aspiration of gastric contents is a complication responsible for the third highest cause of anaesthesia-related mortality in France, and for 50% of airway management-related mortality in the UK. The occurrence of pulmonary aspiration of gastric contents is often the result of a poor assessment of the risk of a "full" stomach, and could therefore often be avoided if the preoperative gastric contents were known to the anaesthetist. It is therefore useful to be able to discriminate easily between patients at risk of aspiration and those at low risk before general anaesthesia, and this can be done by ultrasound examination of the gastric contents in the gastric antrum, non-invasively (abdominal ultrasound) using a 2-5 MHz abdominal ultrasound probe or a high-frequency linear probe in small children (under 10 kg). European recommendations on preoperative fasting in paediatrics recommend that the examination should be interpreted in a qualitative manner only, without measuring the antral surface. However, the diagnostic performance of this qualitative approach alone has never been evaluated. The aim of this study was to determine the diagnostic performance of the qualitative assessment of gastric contents by ultrasound in children, and to compare it with that of the clinical algorithm, for the detection of a volume of fluid greater than 1.25 ml/kg.

Children will present themselves in the morning after fasting. Upon arrival, if their weight is not known, the children will be weighed. Subsequently, they will be positioned on an examination table in a supine inclined position at 45° (head of the bed elevated). An initial gastric ultrasound will be performed by a physician (investigator 1) who will not conduct the study ultrasounds. This initial ultrasound aims to confirm the absence of gastric content in the supine and right lateral decubitus positions, thereby establishing gastric emptiness.

Investigator 1 will then proceed with the random selection of the clear liquid volume to be ingested for the study.

The child will then be asked to drink this determined volume of clear liquid (water or apple juice according to their preference), as per the randomization results, under the supervision of the first investigator who performed the initial ultrasound.

Subsequently, investigator 2 will perform a gastric ultrasound blindly with respect to the ingested liquid volume, three minutes after the consumption of the clear liquid. The examination will last a maximum of 3 minutes.

Non-invasive gastric antrum ultrasound examinations will utilize a probe with a frequency of 2-5.5 MHz and a linear probe with a frequency of 10 MHz, enabling the evaluation of the gastric antrum's appearance. The diameters (longitudinal D1 and anteroposterior D2) of the antrum will also be measured in the supine (semi-seated and lying) and right lateral positions in the sagittal plane passing through the abdominal aorta and the left lobe of the liver, for the calculation of the antral section area, given by the formula: Antral area = π x D1 x D2 / 4.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 1 and 10 years
* Healthy volunteer, with no significant medical history (American Society of Anesthesiologists class ASA 1)
* Fasting according to the 2022 recommendations of the European Society of Anaesthesia: minimum fasting time of 1 h for clear liquids, 3 h for breast milk, 4 h for infant formula, 6 h for solid non-fatty foods and milk, 8 h for richer meals
* Informed consent signed by the child's legal representatives,
* affiliated to a social security scheme

Exclusion Criteria:

* Agitation of the child preventing gastric ultrasound scans from being performed
* Non-compliance with fasting instructions
* Previous oeso-gastro-duodenal surgery
* Treatments affecting gastric motility (erythromycin, metoclopramide, etc.)
* Obesity defined by a body mass index ≥ 30 kg/m².
* Pathologies that may affect gastric volume: insulin-dependent or requiring diabetes, gastro-oesophageal reflux, scleroderma, etc.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the qualitative examination of the gastric antrum for the detection of gastric fluid volume ≥ 1.25 ml/kg in the 45° semirecumbent position | 3 minutes after the ingestion of water
  Calculation of the sensitivity and specificity

SECONDARY OUTCOMES:
Positive predictive value, negative predictive value, positive and negative likelihood ratio of the qualitative examination of the gastric antrum for the detection of gastric fluid volume ≥ 1.25 ml/kg in the 45° semirecumbent position | 3 minutes after the ingestion of water
  Calculation of the positive predictive value, negative predictive value, positive and negative likelihood ratio
Diagnostic performance of a clinical algorithm used for the interpretation of gastric ultrasound for the detection of gastric fluid volume ≥ 1.25 ml/kg in the 45° semirecumbent position | 3 minutes after the ingestion of water
  Calculation of the sensitivity, specificity, positive predictive value, negative predictive value, positive and negative likelihood ratiovalue, positive and negative likelihood ratio

CONTACTS AND LOCATIONS:
Overall Officials: Lionel BOUVET, Dr, Principal Investigator — Hôpital Femme Mère Enfant
Locations (1):
- Hopital Femme Mère Enfant, Bron, France

REFERENCES:
- [Result] Cercueil E, Henriet A, Barbe C, Santos Machado G, Bouvet L. Diagnostic accuracy of qualitative gastric ultrasound assessment for detecting high gastric fluid volume in children: a prospective randomised study. Anaesthesia. 2025 Jun;80(6):636-644. doi: 10.1111/anae.16539. Epub 2025 Jan 7. PMID 39764617